CLINICAL TRIAL: NCT03214666
Title: GTB-3550 (CD16/IL-15/CD33)Tri-Specific Killer Engager (TriKE®) for the Treatment of High Risk Myelodysplastic Syndromes, Refractory/Relapsed Acute Myeloid Leukemia and Advanced Systemic Mastocytosis
Brief Title: GTB-3550 Tri-Specific Killer Engager (TriKE®) for High Risk Hematological Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Development of GTB-3550 halted due to development of the second generation camelid nanobody TriKE drug product, GTB-3650.
Sponsor: GT Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2015LS167; HM2015-39 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: High-risk Myelodysplastic Syndromes; Acute Myelogenous Leukemia; Systemic Mastocytosis; Mast Cell Leukemia
Keywords: Myelodysplastic Syndromes (MDS); Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Mastocytosis, Systemic; Leukemia, Mast-Cell; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GTB-3550 TriKE® (Phase I: Dose Finding Component) (Experimental): Patients receive a single course of GTB-3550 TriKE® at their assigned dose as 3 weekly treatment blocks. Each block consists of four consecutive 24 hour continuous infusions (over approximately 96 hours) of GTB-3550 TriKE® followed by a 72 hour break after Block #1 and #2. All treatment is given as an inpatient. The assigned dose will be calculated on a weight obtained within 5 days prior to or on day of the 1st dose. The dose is not be recalculated for subsequent treatment blocks.
  Interventions: Drug: GTB-3550 TriKE® Phase I
- GTB-3550 TriKE® Only (Phase II: Extended Component) (Experimental): The treatment schedule is identical to the dose finding component. The extended component uses a Simon's MiniMax two-stage design for continued enrollment using the maximum tolerated dose (MTD) established during Phase I with monitoring guidelines to stop the study early for excessive toxicity.
  Interventions: Drug: GTB-3550 TriKE® Phase II

INTERVENTIONS:
Drug: GTB-3550 TriKE® Phase I — The 1st two patients will be assigned Dose Level 1. The study statistician will assign each new cohort of 2 patients to the most appropriate dose level based on updated toxicity probabilities.
  * Dose Level 1 - 5 μg/kg/day
  * Dose Level 2 - 10 μg/kg/day
  * Dose Level 3 - 25 μg/kg/day
  * Dose Level 4 - 50 μg/kg/day
  * Dose Level 5 - 100 μg/kg/day
  * Dose Level 6 - 150 μg/kg/day
  * Dose Level 7 - 200 μg/kg/day
  Other Names: CD16/IL-15/CD33
  Arms: GTB-3550 TriKE® (Phase I: Dose Finding Component)
Drug: GTB-3550 TriKE® Phase II — Patients will receive the maximum tolerated dose (MTD) established during Phase I with monitoring guidelines to stop the study early for excessive toxicity.
  Other Names: CD16/IL-15/CD33
  Arms: GTB-3550 TriKE® Only (Phase II: Extended Component)

SUMMARY:
This is a multi-center Phase I/II clinical trial of GTB-3550 (CD16/IL-15/CD33) tri-specific killer cell engager (TriKE®) for the treatment of CD33-expressing high risk myelodysplastic syndromes, refractory/relapsed acute myeloid leukemia or advanced systemic mastocytosis. The hypothesis is that GTB-3550 TriKE® will induce natural killer cell function by targeting malignant cells as well as CD33+ myeloid derived suppressor cells (MDSC) which contribute to tumor induced immunosuppression. Because CD16 is the most potent activating receptor on natural killer (NK) cells, this single agent may induce a targeted anti-CD33+ tumor response.

ELIGIBILITY:
Inclusion Criteria: Eligible Diseases

* Diagnosis of one of the following CD33-expressing myeloid malignancies with greater than or equal to 50% CD33+ target cells with no good standard of care treatment options including:
* High Risk Myelodysplastic Syndromes (MDS) progressive on two or more prior regimens and requiring treatment that meets at least one of the following:

  * Revised International Prognostic Scoring System (IPSS-R) High or Very High Risks
  * World Health Organization (WHO) Classification: Refractory anemia with excess blasts-1 (RAEB-1) or RAEB-2
  * Poor and very-poor risk cytogenetic abnormality as defined by the IPSS-R cytogenetic classifications
  * WHO Based Prognostic Scoring System (WPSS): High or Very High Risk
* Therapy related MDS and not a candidate for induction chemotherapy or had an inadequate treatment response after induction chemotherapy.
* Refractory or Relapsed Acute Myelogenous Leukemia (AML) meeting at least one of the following:

  * Refractory AML defined as failure to achieve remission after at least 3 induction attempts

    ** Elderly AML not fit for induction therapy can be enrolled after 2 failed inductions
  * Relapsed AML

    * Not a candidate for hematopoietic stem cell transplant (HSCT), at least one re-induction attempt required
    * Prior HSCT relapse beyond 3 months may be included only if off immunosuppression for a minimum of 4 weeks and do not have graft-versus-host disease (GVHD)
* Advanced systemic mastocytosis (defined as mast cell leukemia, aggressive systemic mastocytosis, and systemic mastocytosis associated with hematologic neoplasm) may enroll without any prior treatment, given there is no standard established therapy.

Inclusion Criteria: Age, Performance Status, Organ Function, Contraception Use

* At least 18 years of age
* Karnofsky score ≥ 70%
* Adequate organ function within 14 days (30 days for cardiac and pulmonary) of study enrollment defined as:

  * Renal: an estimated glomerular filtration rate ≥ 60 mL/min/1.73 m2
  * Hepatic: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and total bilirubin within normal range
  * Pulmonary function: Diffusing capacity for carbon monoxide (DLCO) corrected (ml/min/mm Hg) defined as no more than 5 units below lower limit of normal (Common Terminology Criteria for Adverse Events [CTCAE] v5 Grade 1 carbon monoxide diffusing capacity decreased) based on patient's height, weight, and gender as reported by the institutional pulmonary function lab.
  * Cardiac: Absence of decompensated congestive heart failure, or uncontrolled arrhythmia; left ventricular ejection fraction ≥ 45% by echocardiogram, multigated acquisition (MUGA) scan or cardiac MRI.
* Absolute lymphocyte count (ALC) ≥ 200 cells/mm³ OR absolute circulating CD56+/CD3- NK cell count >25 cells/μl within the 14 days prior to start of therapy
* Sexually active females of childbearing potential and males with partners of child-bearing potential must agree to use adequate birth control during study treatment
* Participant provides voluntary written consent signed before performance of any study-related procedure not part of normal medical care

Exclusion Criteria

* New or progressive pulmonary infiltrates on screening chest x-ray or chest computerized tomography (CT) scan unless cleared for study by Pulmonary. Infiltrates attributed to infection must be stable/improving with associated clinical improvement after 1 week of appropriate therapy (4 weeks for presumed or documented fungal infections).
* Uncontrolled bacterial, fungal or viral infections, known history of HIV
* Active Hepatitis B or Hepatitis C (virus detectable by polymerase chain reaction [PCR]) - chronic asymptomatic viral hepatitis is allowed
* Other concurrent active cancer within the last year (excluding non-melanoma skin cancers)
* Severely clinically obese patients, BMI >38
* Currently taking any over-the-counter (OTC), vitamin, mineral, or dietary supplement within 14 days prior to study drug administration on Day 1 and during study conduct that may confound study safety goals (e.g., St. John's wort). Questions should be discussed with GT Biopharma.
* Pregnant or breast feeding. The effect of GTB-3550 TriKE on the fetus is unknown. Females of childbearing potential must have a blood test within 7 days prior to enrollment to rule out pregnancy - must be repeated if not within 7 days of treatment initiation
* History of central nervous system (CNS) malignancy or symptoms of active CNS disease
* A family history of long QT syndrome or with a corrected QT (QTc) interval > 480 msec at screening
* Currently taking medications known to prolong QT/QTc interval as the potential risk of QT/QTc prolongation is unknown in humans.
* A candidate for potentially curative therapy, including hematopoietic cell transplant
* Unwilling to remain within a 90 minute drive of the study center through at least Day 29

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Juckett, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day: Patients receive a single course of GTB-3550 TriKE® at their assigned dose of 5 ug/kg/day as 3 weekly treatment blocks. Each block consisted of four consecutive 24 hour continuous infusions (over approximately 96 hours) of GTB-3550 TriKE® followed by a 72 hour break after Block #1 and #2. All treatment was given as an inpatient. The assigned dose was calculated on a weight obtained within 5 days prior to or on day of the 1st dose. The dose was not recalculated for subsequent treatment blocks.
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day: Patients receive a single course of GTB-3550 TriKE® at their assigned dose of 10 ug/kg/day as 3 weekly treatment blocks. Each block consisted of four consecutive 24 hour continuous infusions (over approximately 96 hours) of GTB-3550 TriKE® followed by a 72 hour break after Block #1 and #2. All treatment was given as an inpatient. The assigned dose was calculated on a weight obtained within 5 days prior to or on day of the 1st dose. The dose was not recalculated for subsequent treatment blocks.
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day: Patients receive a single course of GTB-3550 TriKE® at their assigned dose of 25 ug/kg/day as 3 weekly treatment blocks. Each block consisted of four consecutive 24 hour continuous infusions (over approximately 96 hours) of GTB-3550 TriKE® followed by a 72 hour break after Block #1 and #2. All treatment was given as an inpatient. The assigned dose was calculated on a weight obtained within 5 days prior to or on day of the 1st dose. The dose was not recalculated for subsequent treatment blocks.
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day: Patients receive a single course of GTB-3550 TriKE® at their assigned dose of 50 ug/kg/day as 3 weekly treatment blocks. Each block consisted of four consecutive 24 hour continuous infusions (over approximately 96 hours) of GTB-3550 TriKE® followed by a 72 hour break after Block #1 and #2. All treatment was given as an inpatient. The assigned dose was calculated on a weight obtained within 5 days prior to or on day of the 1st dose. The dose was not recalculated for subsequent treatment blocks.
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day: Patients receive a single course of GTB-3550 TriKE® at their assigned dose of 100 ug/kg/day as 3 weekly treatment blocks. Each block consisted of four consecutive 24 hour continuous infusions (over approximately 96 hours) of GTB-3550 TriKE® followed by a 72 hour break after Block #1 and #2. All treatment was given as an inpatient. The assigned dose was calculated on a weight obtained within 5 days prior to or on day of the 1st dose. The dose was not recalculated for subsequent treatment blocks.
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day: Patients receive a single course of GTB-3550 TriKE® at their assigned dose of 150 ug/kg/day as 3 weekly treatment blocks. Each block consisted of four consecutive 24 hour continuous infusions (over approximately 96 hours) of GTB-3550 TriKE® followed by a 72 hour break after Block #1 and #2. All treatment was given as an inpatient. The assigned dose was calculated on a weight obtained within 5 days prior to or on day of the 1st dose. The dose was not recalculated for subsequent treatment blocks.
Period: Cohort 1: Dose Level 1: 5 ug/kg/Day
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
Started | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2: Dose Level 2: 10ug/kg/Day
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
Started | 0 | 2 | 0 | 0 | 0 | 0
Completed | 0 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 3: Dose Level 3: 25 ug/kg/Day
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
Started | 0 | 0 | 2 | 0 | 0 | 0
Completed | 0 | 0 | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 4: Dose Level 4: 50 ug/kg/Day
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
Started | 0 | 0 | 0 | 2 | 0 | 0
Completed | 0 | 0 | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 5: Dose Level 5: 100 ug/kg/Day
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
Started | 0 | 0 | 0 | 0 | 2 | 0
Completed | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Period: Cohort 6: Dose Level 6: 150 ug/kg/Day
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
Started | 0 | 0 | 0 | 0 | 0 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day: Patients received a single course of GTB-3550 TriKE® at their assigned dose of 5 ug/kg/day as 3 weekly treatment blocks.
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day: Patients received a single course of GTB-3550 TriKE® at their assigned dose of 10 ug/kg/day as 3 weekly treatment blocks.
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day: Patients received a single course of GTB-3550 TriKE® at their assigned dose of 25 ug/kg/day as 3 weekly treatment blocks.
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day: Patients received a single course of GTB-3550 TriKE® at their assigned dose of 50 ug/kg/day as 3 weekly treatment blocks.
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day: Patients received a single course of GTB-3550 TriKE® at their assigned dose of 100 ug/kg/day as 3 weekly treatment blocks.
- GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day: Patients received a single course of GTB-3550 TriKE® at their assigned dose of 150 ug/kg/day as 3 weekly treatment blocks.
- Total: Total of all reporting groups
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 0 | 0 | 0 | 2 | 4
  >=65 years | 1 | 1 | 2 | 2 | 2 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2 | 1 | 1 | 6
  Male | 1 | 1 | 2 | 0 | 1 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 2 | 1 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 2 | 2 | 2 | 12
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 2 | 2 | 2 | 2 | 2
Baseline Disease [Count of Participants; unit: Participants]
  Relapsed/Refractory Acute Myeloid Leukemia (AML) - Secondary AML | 1 | 0 | 1 | 0 | 1 | 1 | 4
  Relapsed/Refractory AML - de novo AML | 1 | 1 | 1 | 0 | 0 | 1 | 4
  Relapsed/Refractory AML - Treatment-related | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Myelodysplastic Syndrome (MDS) | 0 | 1 | 0 | 2 | 0 | 0 | 3
Number of Prior Lines of Cancer Therapy [Count of Participants; unit: Participants] — The number of prior lines of cancer therapies include therapies to treat any cancer diagnosis.
  Participants
    2 | 0 | 0 | 2 | 0 | 0 | 1 | 3
    3 | 1 | 0 | 0 | 2 | 0 | 0 | 3
    4 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    5 | 0 | 1 | 0 | 0 | 0 | 1 | 2
    6 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    7 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    9 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: GTB-3550 Dosing Summary
Description: The study was terminated prior to reaching the maximal tolerated dose. This outcome measure presents information regarding the number of participants receiving each dose of GTB-3550.
Time Frame: Day 1 (start of GTB-3550 therapy)
Measure: Count of Participants; unit: Participants
Groups:
- GTB-3550 TriKE® (Phase I: Dose Finding Component): Patients received a single course of GTB-3550 TriKE® at their assigned dose as 3 weekly treatment blocks. Patients were assigned 1 of 6 dose levels from 5-150 μg/kg/day.
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component)
Number analyzed (Participants) | 12
Participants
  5 ug/kg/day Dose | 2
  10 ug/kg/day Dose | 2
  25 ug/kg/day Dose | 2
  50 ug/kg/day Dose | 2
  100 ug/kg/day Dose | 2
  150 ug/kg/day Dose | 2

2. Primary Outcome: GTB-3550 Extent of Treatment (Summary)
Description: This outcome measure summarizes the number of GTB-3550 treatment blocks participants received during the first cycle of treatment.
Time Frame: Day 28 relative to the start of GTB-3550 therapy
Measure: Count of Participants; unit: Participants
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2
Participants
  Number of Participants Completing Blocks 1-3 | 2 | 2 | 2 | 2 | 1 | 2
  Number of Participants Completing Only Blocks 1 and 2 | 0 | 0 | 0 | 0 | 1 | 0

3. Secondary Outcome: Number of GTB-3550 TriKE® Treatment-Emergent Adverse Events (TEAEs) [Safety and Tolerability]
Description: The number of unexpected events in relation to GTB-3550 TriKE®. TEAEs were measured up to Day 28 relative to GTB-3550 therapy.
Time Frame: Day 28 relative to the start of GTB-3550 therapy
Measure: Number; unit: Events
Units Other Than Participants: TEAEs Regardless of Relationship
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2
Number analyzed (TEAEs Regardless of Relationship) | 62 | 48 | 70 | 28 | 62 | 113
Events
  Unexpected and Related TEAEs | 0 | 0 | 0 | 0 | 0 | 3
  Unexpected and Related Serious Adverse Events | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Number of patients surviving at 6 months post-treatment on this study.
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2
participants | 1 | 0 | 2 | 1 | 1 | 0

5. Secondary Outcome: Number of Participants Experiencing a Reduction in Blast Count Post-GTB-3550 Therapy
Description: Blast count was measured at the time of standard of care disease assessment after GTB-3550 therapy. Blast percent was assessed by morphology and/or flow cytometry.
Time Frame: After Day 28 Relative to GTB-3550 Therapy
Measure: Number; unit: participants
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2
participants | 0 | 0 | 1 | 1 | 1 | 1

6. Post Hoc Outcome: Number of Participants Proceeding to an Optional 2nd Cycle of GTB-3550 Therapy
Description: Participants with lack of disease progression or evidence of a clinical improvement had the opportunity to receive an optional 2nd cycle of therapy ('retreatment').
Time Frame: 2-4 weeks after completion of the 1st cycle of therapy
Measure: Number; unit: participants
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2
participants | 1 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected beginning with the first dose of GTB-3550 (Day 1) through Day 29 after the start of GTB-3550 therapy. All-cause mortality was monitored for up to 6 months after the start of GTB-3550 therapy.
Description: Adverse events were assessed at the following study timepoint: prior to the infusion start of each 24 hour infusion (i.e. Days 1-4, 8-11 and 15-18), at the end of the final infusion of each block (i.e. Days 5, 12, and 19), Day 22 and Day 29.
Arm/Group | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day
All-Cause Mortality (participants affected / at risk) | 1/2 | 2/2 | 0/2 | 1/2 | 1/2 | 2/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 1/2 | 0/2 | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 2/2 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day (N=2) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day (N=2) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day (N=2) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day (N=2) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day (N=2) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) — All Grade 3; 2 possibly related to GTB-3550
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Grade 3; Unlikely related to GTB-3550
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 3; Unrelated to GTB-3550
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 5 ug/kg/Day (N=2) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 10 ug/kg/Day (N=2) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 25 ug/kg/Day (N=2) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 50 ug/kg/Day (N=2) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 100 ug/kg/Day (N=2) | GTB-3550 TriKE® (Phase I: Dose Finding Component): 150 ug/kg/Day (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (12) — Grade 2 count: 5 (2 possibly related to GTB-3550) Grade 3 count: 14 (5 possibly related to GTB-3550)
LDH Increase (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unrelated to GTB-3550)
C-reactive protein increase (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Possibly related to GTB-3550)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 1 (2) | 2 (3) — Grade 3 Count: 10 (6 possibly related to GTB-3550)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Grade 2 Count: 1 (Unrelated to GTB-3550)
Sinus tachycardia (Cardiac disorders) | 1 (3) | 2 (4) | 0 (0) | 1 (1) | 2 (3) | 2 (6) — Grade 1 Count: 15 (9 possibly and 1 probably related to GTB-3550) Grade 2 Count: 2 (2 possibly related to GTB-3550)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 Grade 2 Count: 1 Unrelated to GTB-3550
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 3 (1 possibly related to GTB-3550)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unrelated to GTB-3550)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 2 Count: 1 (Unrelated to GTB-3550)
Gingival bleeding/blood blister (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 2 Count: 1 (Unlikely related to GTB-3550)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 2 Count: 1 (Unrelated to GTB-3550)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Grade 2 Count: 2 Grade 1 Count: 1 Unrelated/unlikely related to GTB-3550
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 1 Count: 1 (Unrelated to GTB-3550)
Chills (General disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 2 (6) — Grade 1 Count: 10 (6 possibly and 3 probably related to GTB-3550) Grade 2 Count: 3 (2 possibly related to GTB-3550)
Edema limbs (General disorders) | 0 (0) | 1 (5) | 1 (1) | 2 (2) | 2 (4) | 1 (1) — Grade 1 Count: 10 (4 possibly related to GTB-3550) Grade 2 Count: 3 (1 possibly related to GTB-3550)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) — Grade 1 Count: 2 (1 possibly related to GTB-3550) Grade 2 Count: 3 (1 possibly related to GTB-3550)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (4) | 2 (14) — Grade 1 Count: 13 (7 possibly and 5 probably related to GTB-3550) Grade 2 Count: 7 (2 possibly and 5 probably related to GTB-3550) Grade 3 Count: 1 (Probably related to GTB-3550)
IL-6 Increase (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unlikely related to GTB-3550)
Chloride increased (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 2 (Unlikely related to GTB-3550)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unlikely related to GTB-3550)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 2 Count: 1 (Unrelated to GTB-3550)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 2 Count: 1 (Unlikely related to GTB-3550)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 1 Count: 2 (1 possibly and 1 probably related to GTB-3550)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 1 Count: Mild (Unlikely related to GTB-3550)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 1 (1) — Grade 1 Count: 4 (1 possibly related to GTB-3550) Grade 2 Count: 2 (2 possibly related to GTB-3550) Grade 3 Count: 2 (2 possibly related to GTB-3550)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2) — Grade 1 Count: 5 (1 possibly and 1 probably related to GTB-3550)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) — Grade 1 Count: 2 (1 possibly related to GTB-3550) Grade 2 Count: 1 (Possibly related to GTB-3550) Grade 3 Count: 2 (2 Possibly related to GTB-3550)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unrelated to GTB-3550)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) — Grade 1 Count: 4 (1 possibly related to GTB-3550)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (3) | 2 (3) | 2 (4) | 2 (8) | 2 (5) — Grade 1 Count: 16 (4 possibly related to GTB-3550) Grade 2 Count: 6 (3 possibly related to GTB-3550) Grade 3 Count: 1 (unrelated to GTB-3550)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (unrelated to GTB-3550)
IL-6 increase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Possibly related to GTB-3550)
LDH elevated - intermittent (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (unrelated to GTB-3550)
Ferritin elevation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (unrelated to GTB-3550)
CRP elevation (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 3 (1 probably related to GTB-3550)
Fibrinogen elevation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (unrelated to GTB-3550)
Chloride increase - intermittent (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 2 (Unrelated to GTB-3550)
Lymphocyte count decreased (Investigations) | 1 (2) | 2 (2) | 2 (7) | 1 (3) | 2 (6) | 1 (4) — Grade 1 Count: 2 (2 probably related to GTB-3550) Grade 2 Count: 9 (1 possibly and 6 probably related to GTB-3550) Grade 3 Count: 10 (1 possibly and 5 possibly related to GTB-3550) Grade 4 Count: 3 (3 probably related to GTB-3550)
Neutrophil count decreased (Investigations) | 1 (5) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) — Grade 2 Count: 2 (2 possibly related to GTB-3550) Grade 3 Count: 2 (1 possibly related to GTB-3550) Grade 4 Count: 9 (1 possibly related to GTB-3550)
Platelet count decreased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (7) — Grade 3 Count: 4 (unrelated to GTB-3550) Grade 4 Count: 11 (unrelated or unlikely related to GTB-3550)
White blood cell decreased (Investigations) | 1 (5) | 1 (1) | 1 (3) | 1 (4) | 2 (2) | 1 (4) — Grade 1 Count: 1 (Probably related to GTB-3550) Grade 2 Count: 1 (Possibly related to GTB-3550) Grade 3 Count: 7 (3 possibly related to GTB-3550) Grade 4 Count: 10 (5 possibly and 2 probably related to GTB-3550)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 1 Count: 1 (Unlikely related to GTB-3550) Grade 3 Count: 1 (Unrelated to GTB-3550)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unlikely related to GTB-3550)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) — Grade 1 Count: 4 (Unrelated or unlikely related to GTB-3550)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unlikely related to GTB-3550)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | 2 (2) | 2 (13) | 1 (1) | 2 (3) | 1 (1) — Grade 1 Count: 16 (1 possibly related to GTB-3550) Grade 2 Count: 8 (Unrelated or unlikely related to GTB-3550)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 1 (3) | 1 (4) — Grade 1 Count: 8 (2 possibly related to GTB-3550) Grade 2 Count: 4 (Unlikely related to GTB-3550) Grade 3 Count: 1 (Unrelated to GTB-3550)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) — Grade 1 Count: 1 (Unlikely related to GTB-3550) Grade 2 Count: 3 (1 possibly and 1 probably related to GTB-3550)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unrelated to GTB-3550)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unrelated to GTB-3550)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) — Grade 1 Count: 1 (Possibly related to GTB-3550) Grade 2 Count: 2 (1 Possibly related to GTB-3550)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 2 Count: 1 (Unlikely related to GTB-3550)
Muscle spasms, intermittent (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 2 Count: 1 (Unlikely related to GTB-3550)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 2 Count: 2 (Unrelated to GTB-3550)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 2 Count: 3 (Unrelated or unlikely related to GTB-3550)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 1 Count: 1 (Possibly related to GTB-3550)
Headache (Nervous system disorders) | 1 (3) | 1 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (2) — Grade 1 Count: 10 (2 possibly related to GTB-3550) Grade 2 Count: 1 (Unlikely related to GTB-3550)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 2 Count: 1 (Unlikely related to GTB-3550)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unrelated to GTB-3550)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 2 Count: 1 (Unrelated to GTB-3550)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unrelated to GTB-3550)
Restlesness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unlikely related to GTB-3550)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Grade 2 Count: 1 (Unrelated to GTB-3550)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 1 Count: 1 (Unlikely related to GTB-3550)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 2 (Unrelated or unlikely related to GTB-3550)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (2) — Grade 1 Count: 5 (3 possibly related to GTB-3550) Grade 2 Count: 1 (Unlikely related to GTB-3550) Grade 3 Count: 1 (Unlikely related to GTB-3550)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 2 (4) — Grade 1 Count: 3 (2 possibly related to GTB-3550) Grade 2 Count: 5 (3 possibly related to GTB-3550) Grade 3 Count: 1 (Unlikely related to GTB-3550)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 2 Count: 1 (Unlikely related to GTB-3550)
On oxygen with no documented hypoxia, intermittent (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 2 Count: 1 (Possibly related to GTB-3550)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unlikely related to GTB-3550)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) — Grade 1 Count: 1 (Unrelated to GTB-3550) Grade 2 Count: 1 (Unlikely related to GTB-3550) Grade 3 Count: 1 (Unlikely related to GTB-3550)
Rash - L leg (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 1 Count: 1 (Unrelated to GTB-3550)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 1 Count: 1 (Possibly related to GTB-3550)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 2 (2) | 2 (2) — Grade 1 Count: 3 (1 possibly related to GTB-3550) Grade 2 Count: 4 (Unrelated or unlikely related to GTB-3550) Grade 3 Count: 4 (Unrelated to GTB-3550)
Hypotension (Vascular disorders) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (7) — Grade 1 Count: 9 (8 possibly and 1 probably related to GTB-3550) Grade 2 Count: 3 (3 possibly related to GTB-3550)

LIMITATIONS AND CAVEATS:
This trial was terminated due to plans to clinically advance a modified second generation TriKE, requiring a new phase 1 study. Given this early termination, the maximal tolerated dose was not reached and the study did not proceed to phase 2. As only 12 participants were enrolled, the outcomes are presented in summary/descriptive format only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT03214666/Prot_SAP_000.pdf